CLINICAL TRIAL: NCT03512262
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Multicenter Study to Evaluate the Safety and Efficacy of Abaloparatide-SC for the Treatment of Men With Osteoporosis
Brief Title: Safety and Efficacy of Abaloparatide-SC in Men With Osteoporosis (ATOM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BA058-05-019; ATOM (Other: Radius Health, Inc.)
Record Dates: First submitted 2018-04-17; First posted 2018-04-30 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Osteoporosis; Osteoporosis, Age-Related; Osteoporosis Localized to Spine; Age Related Osteoporosis; Osteoporosis Senile; Osteoporosis of Vertebrae
Keywords: BA058; abaloparatide; abaloparatide-SC; osteoporosis; male osteoporosis; TYMLOS®; fracture; bone loss
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; Bone Diseases, Metabolic | interventions — abaloparatide

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 treatment ratio (abaloparatide:placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment will be blinded to participants, investigators, outcome Assessor and care provider throughout the study except in a medical emergency where the identity of study medication is necessary to appropriately treat the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abaloparatide (Experimental): Participants self-administered daily doses of abaloparatide 80 mcg SC using a single-participant, multiple-use, prefilled injection pen that delivers 30 doses. Participants received a new injection pen every 30 days.
  Interventions: Drug: Abaloparatide
- Placebo (Placebo Comparator): Participants self-administered daily doses of placebo SC using a single-participant, multiple-use, prefilled injection pen that delivers 30 doses. Participants received a new injection pen every 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abaloparatide — Abaloparatide is a synthetic peptide that is a potent and selective activator of the parathyroid hormone 1 receptor signaling pathway.
  Other Names: TYMLOS®; BA058; abaloparatide-SC
  Arms: Abaloparatide
Drug: Placebo — Abaloparatide-matched placebo.
  Arms: Placebo

SUMMARY:
A 12-month study to measure the efficacy and safety of abaloparatide in men with osteoporosis.

DETAILED DESCRIPTION:
The primary objective of this prospective controlled study is to evaluate the efficacy and the safety of abaloparatide 80 micrograms (mcg) per day administered subcutaneously (SC) compared to placebo in men with osteoporosis. Efficacy was primarily assessed by the change in bone mineral density (BMD) over 12 months.

ELIGIBILITY:
Key Inclusion Criteria

* Healthy ambulatory male from 40 to 85 years of age (inclusive) with primary osteoporosis or osteoporosis associated with hypogonadism.
* The participant has a BMD T-score based on female or male reference range (depending on date of enrollment) as assessed by the central imaging vendor of ≤ -2.5 at the lumbar spine (L1-L4) or hip (femoral neck or total hip) by dual energy X-ray absorptiometry (DXA) or ≤ -1.5 and with radiologic evidence of vertebral fracture or a documented history of low-trauma nonvertebral fracture sustained in the past 5 years. Men older than 65 years may be enrolled if they have a BMD T-score ≤ -2.0 even if they do not meet the fracture criteria.
* Normal medical history, physical examination, including vital signs, and body mass index.
* Hypogonadal participants whose doses of androgens have been stable for at least twelve months before randomization are eligible and may continue therapy during the study.
* Laboratory tests within the normal range including serum calcium (albumin-corrected), parathyroid hormone, serum phosphorus and alkaline phosphatase, and thyroid stimulating hormone values.

Key Exclusion Criteria

* Presence of abnormalities of the lumbar spine that would prohibit assessment of spinal BMD, defined as having at least 2 radiologically evaluable vertebrae within L1-L4.
* A BMD T-score of ≤-3.5 at the total hip, femoral neck, or lumbar spine based on female or male reference range (depending on date of enrollment).
* Unevaluable hip BMD or participants who have undergone bilateral hip replacement.
* Fragility fracture within the prior twelve months.
* History of severe vertebral fracture or >2 moderate vertebral fractures.
* History of bone disorders (for example, Paget's disease) other than osteoporosis.
* participant with clinical signs of hypogonadism present at screening who plan to initiate testosterone replacement.
* History of prior external beam or implant radiation therapy involving the skeleton other than radioiodine.
* History of chronic or recurrent renal, hepatic, pulmonary, allergic, cardiovascular, gastrointestinal, endocrine, central nervous system, hematologic or metabolic diseases, or immunologic, emotional and/or psychiatric disturbances to a degree that would interfere with the interpretation of study data or compromise the safety of the participant.
* History of Cushing's disease, growth hormone deficiency or excess, hyperthyroidism, hypo- or hyperparathyroidism or malabsorptive syndromes within the past year.

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Marin Endocrine Care & Research, Inc., Greenbrae, California
  - Alta California Medical Group, Simi Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Panorama Orthopedics & Spine Center, Golden, Colorado
  - MedStar Georgetown-MedStar Georgetown Transplant Institute University Hospital (MGUH), Washington D.C., District of Columbia
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Baptist Diabetes Associates, Pa, Miami, Florida
  - Center For Advanced Research & Education, Gainesville, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - SUNY Upstate Medical University, Syracuse, New York
  - PMG Research of Cary, LLC, Cary, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Centex Studies, Inc., Houston, Texas
  - Centex Studies, Inc, McAllen, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - University of Wisconsin Osteoporosis Clinical Research Program, Madison, Wisconsin
- Italy (3):
  - Azienda ospedaliera universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera Universitaria Senese-Policlincio Santa Maria Alle Scotte, Siena, Tuscany
  - Azienda ospedaliera universitaria integrata di verona(AOUI), Verona
- Poland (9):
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - Zdrowie Osteo-Medic s.c. Lidia I Artur Racewicz, Agnieszka I Jerzy Supronik, Bialystok, Podlaskie Voivodeship
  - ClinicMed Daniluk, Nowak Sp.j., Bialystok
  - Centrum Leczenia Osteoporozy Klinika Zdrowej Kosci, Lodz
  - ETG Siedlce, Siedlce
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - NZOZ Nasz Lekarz, Torun
  - Synexus Polska Sp z o.o Oddzial we Wroclawiu, Wroclaw

REFERENCES:
- [Background] Rizzoli R, Bonjour JP, Ferrari SL. Osteoporosis, genetics and hormones. J Mol Endocrinol. 2001 Apr;26(2):79-94. doi: 10.1677/jme.0.0260079. PMID 11241160
- [Background] Mannstadt M, Juppner H, Gardella TJ. Receptors for PTH and PTHrP: their biological importance and functional properties. Am J Physiol. 1999 Nov;277(5):F665-75. doi: 10.1152/ajprenal.1999.277.5.F665. PMID 10564229
- [Background] Dempster DW, Cosman F, Parisien M, Shen V, Lindsay R. Anabolic actions of parathyroid hormone on bone. Endocr Rev. 1993 Dec;14(6):690-709. doi: 10.1210/edrv-14-6-690. No abstract available. PMID 8119233

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who remained eligible for study participation were randomly allocated, using a 2:1 randomization ratio (abaloparatide:placebo) on Day 1, to receive treatment with either blinded abaloparatide 80 micrograms (mcg) per day or daily placebo subcutaneous (SC) injections.
Groups:
- Abaloparatide: Participants self-administered daily doses of abaloparatide 80 mcg SC using a single-participant, multiple-use, prefilled injection pen.
- Placebo: Participants self-administered daily doses of placebo SC using a single-participant, multiple-use, prefilled injection pen.
Period: Overall Study
Arm/Group | Abaloparatide | Placebo
Started | 149 | 79
Received at Least 1 Dose of Study Drug | 149 | 79
Completed | 114 | 64
Not Completed | 35 | 15
Not completed — Adverse Event | 8 | 3
Not completed — Death (non-treatment emergent) | 1 | 0
Not completed — Withdrawal by Subject | 17 | 9
Not completed — Lost to Follow-up | 7 | 1
Not completed — Other than Specified | 2 | 2

BASELINE CHARACTERISTICS:
Population: ITT Population: All participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abaloparatide | Placebo | Total
Number analyzed (Participants) | 149 | 79 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (8.25) | 67.8 (8.53) | 68.3 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 149 | 79 | 228
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 140 | 76 | 216
  Race: Black or African American | 0 | 1 | 1
  Race: Asian | 8 | 1 | 9
  Race: Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Race: Other | 0 | 1 | 1
  Ethnicity: Hispanic or Latino | 23 | 13 | 36
  Ethnicity: Not Hispanic or Latino | 124 | 66 | 190
  Ethnicity: Unknown | 1 | 0 | 1
  Ethnicity: MIssing | 1 | 0 | 1
Lumbar Spine Bone Mineral Density (BMD) T-score [Mean (Standard Deviation); unit: BMD T-Score] — The bone mineral density (BMD) T-score is the BMD, assessed by dual energy x-ray absorptiometry (DXA), at the site when compared to that of a healthy man/woman (20 to 29 years old). Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a man/woman (20 to 29 years old). Lower T-scores indicate worse bone condition.
  BMD T-Score | -2.11 (1.119) | -2.05 (1.217) | -2.09 (1.152)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 12
Description: Lumbar Spine BMD was assessed by DXA scans evaluated by a central imaging laboratory. Lumbar spine scans included L1 through L4. Positive changes from baseline indicate improvement in bone health.
Time Frame: Baseline, Month 12
Population: Intent-to-Treat (ITT) Population: All participants randomized into the study. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 119 | 66
percent change | 8.4820 (0.5353) | 1.1654 (0.7235)
Statistical Analysis 1: Comparison: Abaloparatide vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Significance level of 0.01; Missing values were imputed using a multiple imputation method; Least Squares (LSM) Means Difference = 7.3165, 99% CI 2-sided [5.0668 to 9.5663]

2. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 12
Description: Total hip BMD was assessed by DXA scans evaluated by a central imaging laboratory. Positive changes from baseline indicate improvement in bone health.
Time Frame: Baseline, Month 12
Population: ITT Population: All participants randomized into the study. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 119 | 66
percent change | 2.1351 (0.2711) | 0.0143 (0.3543)
Statistical Analysis 1: Comparison: Abaloparatide vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Significance level of 0.01; Missing values were imputed using a multiple imputation method; LSM Difference = 2.1209, 99% CI 2-sided [0.9948 to 3.2469]

3. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Month 12
Description: Femoral neck BMD was assessed by DXA scans evaluated by a central imaging laboratory. Positive changes from baseline indicate improvement in bone health.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 119 | 66
percent change | 2.9766 (0.3448) | 0.1545 (0.4527)
Statistical Analysis 1: Comparison: Abaloparatide vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Significance level of 0.01; Missing values were imputed using a multiple imputation method; LSM Difference = 2.8221, 99% CI 2-sided [1.3972 to 4.2471]

4. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 6
Description: as for outcome 1
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 123 | 70
percent change | 5.5436 (0.4127) | 0.6418 (0.5472)

5. Secondary Outcome: Percent Change in Total Hip BMD From Baseline at Month 6
Description: as for outcome 2
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 122 | 70
percent change | 1.3888 (0.2142) | 0.0267 (0.2790)

6. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Month 6
Description: as for outcome 3
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 122 | 70
percent change | 1.4790 (0.2714) | -0.1884 (0.3569)

7. Secondary Outcome: Percent Change From Baseline in Ultra-Distal Radius BMD at Month 12
Description: Ultra-distal radius BMD was assessed by DXA scans. Positive changes from baseline indicate improvement in bone health.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 115 | 61
percent change | 1.4358 (0.4236) | -0.1915 (0.5722)

8. Secondary Outcome: Percent Change From Baseline in Distal One-third Radius BMD at Month 12
Description: Distal one-third radius BMD was assessed by DXA scans. Positive changes from baseline indicate improvement in bone health.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 115 | 61
percent change | -0.0138 (0.3253) | 0.7066 (0.4285)

9. Secondary Outcome: Percent Change From Baseline in Serum Procollagen Type I N-terminal Propeptide (s-PINP) at Month 12
Description: Blood samples were taken to measure s-PINP, a bone formation marker. s-PINP concentrations reflect the rate of skeletal new bone formation. Increases in s-PINP indicate anabolic biologic response in the bone.
Time Frame: Baseline, Month 12
Population: ITT Population: All participants randomized into the study. Here, overall number of participants analyzed is the total number of participants who had s-PINP evaluation at Baseline and Month 12.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 119 | 65
percent change | 225.919 (416.4173) | 0.291 (31.8038)

10. Secondary Outcome: Percent Change From Baseline in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) at Month 12
Description: Blood samples were taken to measure s-CTX. Elevated levels of s-CTX indicate increased bone resorption (bone loss).
Time Frame: Baseline, Month 12
Population: ITT Population: All participants randomized into the study. Here, overall number of participants analyzed is the total number of participants who had s-CTX evaluation at Baseline and Month 12.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 119 | 65
percent change | 89.639 (206.7227) | 15.359 (40.3351)

11. Secondary Outcome: Number of Participants With New Clinical Fractures
Description: Radiological evaluations were performed to identify any new clinical fractures (occurring after the screening visit).
Time Frame: Baseline through Month 12
Population: ITT Population: All participants randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 149 | 79
Participants | 1 | 3

12. Secondary Outcome: Percent of Participants With Change in Disease Status
Description: The percentage of participants converting from the categories of osteoporosis to osteopenia or from osteopenia to normal at End of Treatment (Month 12) was assessed. Osteoporosis was defined as lumbar spine or total hip BMD T-score ≤ -2.5. Osteopenia was defined as one of the following:
  * Lumbar spine > -2.5 and total hip BMD T-score > -2.5 and < -1.0
  * Lumbar spine > -2.5 and < -1.0 and total hip BMD T-score > -2.5
  * Normal was defined as lumbar spine and total hip BMD T-score ≥ -1.0.
Time Frame: Baseline through Month 12
Population: ITT Population: All participants randomized into the study. Here, overall number of participants analyzed is the total number of participants who had baseline evaluation and also had end of treatment BMD disease category evaluation (normal, osteopenia, and osteoporosis).
  .
Measure: Number; unit: percentage of participants
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 142 | 75
percentage of participants
  Osteopenia to Normal: number analyzed (Participants) | 68 | 25
  Osteopenia to Normal | 8.8 | 8.0
  Osteopenia to Osteoporosis: number analyzed (Participants) | 68 | 25
  Osteopenia to Osteoporosis | 0 | 12.0
  Osteoporosis to Normal: number analyzed (Participants) | 70 | 47
  Osteoporosis to Normal | 2.9 | 0
  Osteoporosis to Osteopenia: number analyzed (Participants) | 70 | 47
  Osteoporosis to Osteopenia | 57.1 | 12.8
  Normal to Osteopenia or Osteoporosis: number analyzed (Participants) | 4 | 3
  Normal to Osteopenia or Osteoporosis | 0 | 0

13. Secondary Outcome: Percent of Participants Experiencing BMD Gains From Baseline of > 0%, > 3%, and > 6% at the Lumbar Spine, Femoral Neck, and Total Hip
Description: Lumbar spine, femoral neck, and total hip BMD were assessed by DXA scans evaluated by a central imaging laboratory.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 119 | 66
percentage of participants
  BMD Increase >0% at All Three Sites | 67.2 | 15.2
  BMD Increase >3% at All Three Sites | 31.9 | 1.5
  BMD Increase >6% at All Three Sites | 9.2 | 0.0

14. Secondary Outcome: Percent Change From Baseline in Total Hip Volumetric BMD as Measured by Quantitative Computed Tomography (QCT) at Month 12
Description: QCT scans were evaluated by a central imaging laboratory.
Time Frame: Baseline, Month 12
Population: Only 2 participants per reporting group had volumetric BMD measured by QCT at baseline and Month 12, therefore, no data is reported here to maintain participant confidentiality.
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percent Change From Baseline in Femoral Neck Volumetric BMD as Measured by QCT at Month 12
Description: QCT scans were evaluated by a central imaging laboratory.
Time Frame: Baseline, Month 12
Population: as for outcome 14
Arm/Group | Abaloparatide | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Month 13
Description: Safety Population was used for analyses of treatment-emergent serious and "other" adverse events that occurred from Day 1 (after dosing) through Month 13. The one death recorded under "All-cause mortality" was due to an event that was not treatment-emergent.
Arm/Group | Abaloparatide | Placebo
All-Cause Mortality (participants affected / at risk) | 1/149 | 0/79
Serious Adverse Events (participants affected / at risk) | 8/149 | 4/79
Other Adverse Events (participants affected / at risk) | 73/149 | 29/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abaloparatide (N=149) | Placebo (N=79)
Angina unstable (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Skin graft rejection (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Peripheral nerve palsy (Nervous system disorders) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abaloparatide (N=149) | Placebo (N=79)
Injection site erythema (General disorders) | 19 | 4
Injection site swelling (General disorders) | 10 | 0
Injection site pain (General disorders) | 9 | 0
Nasopharyngitis (Infections and infestations) | 13 | 6
Bronchitis (Infections and infestations) | 8 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Sinusitis (Infections and infestations) | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Dizziness (Nervous system disorders) | 13 | 1
Headache (Nervous system disorders) | 8 | 4
Hypertension (Vascular disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT03512262/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT03512262/SAP_001.pdf